CLINICAL TRIAL: NCT00001086
Title: A Randomized, Phase II, Placebo Controlled Trial of Abacavir (ABC, 1592U89) in Combination With Open-Label Indinavir Sulfate (IDV) and Efavirenz (EFV, DMP-266) in HIV-Infected Subjects With Nucleoside Analog Experience: A Rollover Study for ACTG 320
Brief Title: A Study of Abacavir Plus Indinavir Sulfate Plus Efavirenz in HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 368; 11331 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Placebos; HIV-1; Drug Therapy, Combination; HIV Protease Inhibitors; Indinavir; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; abacavir; efavirenz

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Abacavir sulfate
Drug: Efavirenz

SUMMARY:
To compare the virologic response between abacavir (ABC, 1592U89) regimens (drug vs. placebo) and between the 2 dosing regimens (BID vs. TID) with respect to the proportion of patients with plasma HIV RNA levels below the limit of detection [AS PER AMENDMENT 8/27/97: < 500 copies/ml at week 16]. To evaluate the safety and tolerance of the study arms. [AS PER AMENDMENT 3/10/99: During the extension period, compare the time to detectable viremia (2 consecutive plasma HIV RNA levels greater than or equal to 500 copies/ml) between ABC and placebo.] Therapeutically, there is a need to explore potent alternative therapy for patients who have received, or are currently receiving, a double nucleoside analog combination including lamivudine (3TC), a regimen that was proven to be clinically inferior to indinavir (IDV) when combined with zidovudine/3TC in study ACTG 320. In order to produce and maintain a maximal antiviral response, all patients in this study will receive 2 or 3 potent, new agents; ABC, a nucleoside analog, EFV, a non-nucleoside reverse transcriptase inhibitor (NNRTI), and IDV, a protease inhibitor. Virologically, the major question this protocol seeks to answer is how prior 3TC exposure in a dual nucleoside regimen influences the response to subsequent treatment. It is unclear whether it is best to add a protease inhibitor either 1) an NNRTI at 1 of 2 doses, or 2) an NNRTI at 1 of 2 doses plus a new nucleoside analog to achieve plasma HIV RNA levels that are below the limits of detection.

DETAILED DESCRIPTION:
Therapeutically, there is a need to explore potent alternative therapy for patients who have received, or are currently receiving, a double nucleoside analog combination including lamivudine (3TC), a regimen that was proven to be clinically inferior to indinavir (IDV) when combined with zidovudine/3TC in study ACTG 320. In order to produce and maintain a maximal antiviral response, all patients in this study will receive 2 or 3 potent, new agents; ABC, a nucleoside analog, EFV, a non-nucleoside reverse transcriptase inhibitor (NNRTI), and IDV, a protease inhibitor. Virologically, the major question this protocol seeks to answer is how prior 3TC exposure in a dual nucleoside regimen influences the response to subsequent treatment. It is unclear whether it is best to add a protease inhibitor either 1) an NNRTI at 1 of 2 doses, or 2) an NNRTI at 1 of 2 doses plus a new nucleoside analog to achieve plasma HIV RNA levels that are below the limits of detection.

Prior to randomization, patients are stratified by CD4 cell count (cells/mm3): less than or equal to 50 versus greater than 50 and by ACTG 320 participation: enrolled versus not enrolled. Patients with greater than 50 CD4 cells/mm3 are randomized to 1 of 4 treatment arms (Arms I, II, III, or IV) and patients with less than or equal to 50 CD4 cells/mm3 are randomized to 1 of 2 treatment arms (Arms I and II). All patients will be followed for 48 weeks beyond the enrollment of the last patient. The regimens for the treatment arms are as follows: Arm I - indinavir (IDV) plus EFV plus ABC placebo bid, Arm II - IDV (higher dose) plus EFV (lower dose) plus ABC, Arm III - IDV plus EFV plus ABC placebo, and Arm IV - IDV (higher dose) plus EFV (lower dose) plus ABC. If 15 week data indicates this is a reasonable dosing regimen, the sample size in Arms III and IV will be expanded to include additional patients with a CD4 count greater than 50 cells/mm3 and allow for equal enrollment across all 4 treatment arms. Those patients who roll over from ACTG 320 will be assigned to receive open-label treatment on Arm II and evaluated independently of the 4 treatment arms listed above.

[AS PER AMENDMENT 8/27/97: Patients with 2 consecutive HIV RNA measurements at least 500 copies/ml at week 16 or anytime thereafter are given the option to receive open-label treatment with IDV plus EFV plus ABC, or to seek the best available therapy outside of the study. NOTE: Patients who choose the open-label combination may take other prescribed nucleoside analogs provided outside the study.] [AS PER AMENDMENT 12/17/97: It is strongly recommended that patients who reach a confirmed endpoint and elect to receive open-label therapy consider adding additional approved (and novel, if possible) antiretroviral agents to their open-label regimen.] [AS PER AMENDMENT 1/12/98: Patients who choose the open-label combination may receive other approved antiretrovirals obtained outside the study provided the ACTG 368 team approves the combination.] [AS PER AMENDMENT 8/7/98: Subjects will take study medications for a maximum of 96 weeks, depending on their time of study enrollment.] [AS PER AMENDMENT 3/10/99: A 24-week extension, which will end July 30, 1999, has been added to the study. The extension applies to subjects currently on blinded Step 1 treatment, on open-labeled Step 2, or on study but off treatment. Subjects are to be unblinded in their study treatment and followed for the remainder of the extension. Subjects continue on their current study drug schedule. Subjects on blinded IDV plus EFV who, upon unblinding (not failure) decide to add prescription ABC to their regimen, will be considered off study treatment and will be followed for the duration of the extension; those already registered on Step 2 will continue their Step 2 therapy. Any subject who does not wish to continue on the study extension will be unblinded to their original randomized regimen. Subjects who experience virologic failure during the extension should seek best available treatment following current recommendations to use as many approved, novel antiretroviral agents as possible. The new drug regimen may incorporate any or all of the study drugs.]

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Chemoprophylaxis for Pneumocystis carinii pneumonia is required for all patients who have a CD4 cell count <= 200 cells/mm3.
* Topical and/or oral antifungal agents are permitted except for oral ketoconazole.
* Treatment, maintenance or chemoprophylaxis with approved agents for opportunistic infections as clinically indicated, except for rifabutin.
* All antibiotics as clinically indicated.
* Systemic corticosteroid use for <= 21 days for acute problems is permitted as medically indicated; chronic systemic corticosteroid use is not permitted, unless it is within physiologic replacement levels.
* Recombinant erythropoietin and granulocyte colony-stimulating factor are permitted as medically indicated.
* Regularly prescribed medications such as antipyretics, analgesics, allergy medications (except for terfenadine (Seldane) and astemizole (Hismanal)), antidepressants, sleep medications, oral contraceptives, megestrol acetate, testosterone or any other medications are permitted as medically indicated.

NOTE:

* Due to the possibility that EFV or ABC may alter the effectiveness of oral contraceptives or depo-progesterone, oral contraceptives or depo-progesterone must not be used as the sole form of birth control. [AS PER AMENDMENT 8/7/98: adequate birth control is hormonal plus barrier method or two barrier methods].
* Alternative therapies such as vitamins, acupuncture, and visualization techniques will be permitted. Herbal medications should be avoided. Patients should report the use of these therapies; alternative therapies will be recorded. [AS PER AMENDMENT 8/7/98: Due to the likelihood of IDV increasing the concentrations of sildenafil (Viagra) when coadministered, it is suggested that subjects who use viagra take the lowest dose (25 mg, i.e., half the typical dose).]

Both NIAID ACTG 320 participants and non-ACTG 320 patients must have:

* Documented HIV-1 infection.
* Written informed consent from parent or legal guardian for those patients < 18 years old.

Non-ACTG 320 patients must have:

* Documented CD4 cell count <= 200 cells/mm3 at the time of initiation of ZDV (or d4T) plus 3TC therapy [AS PER AMENDMENT 12/17/97:
* Documented CD4 cell count <= 250 cells/mm3 within 3 months of initiation of ZDV (or d4T) plus 3TC therapy].

Prior Medication:

Required:

For ACTG 320 patients:

* Patients must have participated in ACTG 320 with original randomization to the double-nucleoside combination arm, and maintenance of that treatment (on-study/on-treatment in ACTG 320) until enrollment into ACTG 368.

For non-ACTG 320 patients:

* Greater than or equal to 3 months [2 months AS PER AMENDMENT 12/17/97] of therapy with ZDV (or d4T) + 3TC and receiving ZDV (or d4T) + 3TC at the time of entry.

Exclusion Criteria

Co-existing Condition:

Non-ACTG 320 patients with the following symptoms and conditions are excluded:

Malignancy that requires systemic therapy other than minimal Kaposi's sarcoma.

NOTE:

* Minimal Kaposi's sarcoma, defined as <= 5 cutaneous lesions and no visceral disease or tumor-associated edema, allowed, provided systemic therapy not required.

Non-ACTG 320 patients with the following prior conditions or symptoms are excluded:

* Unexplained temperature > 38.5 degrees C for 7 consecutive days.
* Chronic diarrhea defined as > 3 liquid stools per day persisting for 15 days, within 30 days prior to entry.
* Proven or suspected acute hepatitis within 30 days prior to entry, even if AST (SGOT) and ALT (SGPT) are <= 5 X ULN.

Concurrent Medication: Excluded:

* All antiretroviral therapies other then study medications.
* Rifabutin and rifampin.
* Investigational drugs without specific approval from the protocol chair.
* Systemic cytotoxic chemotherapy.
* Oral ketoconazole (Nizoral), terfenadine (Seldane), astemizole (Hismanal), cisapride (Propulsid), triazolam (Halcion), and midazolam (Versed).
* Caution should be taken in the consumption of alcoholic beverages with study medications.
* Itraconazole.

Prior Medication: Excluded: For ACTG 320 patients:

* Those who opted to receive open-label IDV while on ACTG 320, or if they switched to open label IDV during the study.

For non-ACTG 320 patients:

* Acute therapy for an infection or other medical illness within 14 days prior to entry.
* Prior protease inhibitor therapy.
* Prior NNRTI therapy (approved or experimental).
* Erythropoietin, G-CSF or GM-CSF within 30 days prior to entry.
* Interferons, interleukins or HIV vaccines within 30 days prior to entry.
* Any experimental therapy within 30 days prior to entry.
* Rifampin or rifabutin within 14 days prior to entry.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Study Completion 1999-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Squires KE, Study Chair; Hammer SM, Study Chair; Fischl MA, Study Chair
Locations (56):
- United States (55):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - San Francisco Gen Hosp, San Francisco, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Georgetown Univ Hosp, Washington D.C., District of Columbia
  - Howard Univ, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Louis A Weiss Memorial Hosp, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Univ of Iowa Hosp and Clinic, Iowa City, Iowa
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Tulane Med Ctr Hosp, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - State of MD Div of Corrections / Johns Hopkins Univ Hosp, Baltimore, Maryland
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Hennepin County Med Clinic, Minneapolis, Minnesota
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Paul Ramsey Med Ctr, Saint Paul, Minnesota
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Saint Clare's Hosp and Health Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - St Vincent's Hosp / Mem Sloan-Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Moses H Cone Memorial Hosp, Greensboro, North Carolina
  - Central Prison/Women's Prison in Raleigh / NC, Raleigh, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Univ of Kentucky Lexington, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Tennessee / E Tennessee Comprehensive Hemophilia Ctr, Knoxville, Tennessee
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Univ of Texas Galveston, Galveston, Texas
  - Univ of Washington, Seattle, Washington
  - Great Lakes Hemophilia Foundation, Wauwatosa, Wisconsin
- Univ of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Squires K, Hammer S, Degruttola V, Fischl M, Grimes J, Demeter L, Morse G. Randomized trial of abacavir (ABC) in combination with indinavir (IDV) and efavirenz (EFV) in HIV-infected patients (pts) with nucleoside analog experience (NRTI exp). Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:207 (abstract no LB15)
- [Background] Dicenzo R, Forrest A, Smith P, Squires K, Hammer S, Fischl M, Degruttola V, Morse G. Comparing intensive and sparse sampling for estimating the population pharmacokinetics (PK) of indinavir (IDV) in efavirenz (EFV)containing regimens. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 751)
- [Background] Landay AL, Bettendorf D, Chan E, Spritzler J, Schmitz JL, Bucy RP, Gonzalez CJ, Schnizlein-Bick CT, Evans T, Squires KE, Phair JP. Evidence of immune reconstitution in antiretroviral drug-experienced patients with advanced HIV disease. AIDS Res Hum Retroviruses. 2002 Jan 20;18(2):95-102. doi: 10.1089/08892220252779638. PMID 11839142
- [Result] Demeter LM, DeGruttola V, Lustgarten S, Bettendorf D, Fischl M, Eshleman S, Spreen W, Nguyen BY, Koval CE, Eron JJ, Hammer S, Squires K. Association of efavirenz hypersusceptibility with virologic response in ACTG 368, a randomized trial of abacavir (ABC) in combination with efavirenz (EFV) and indinavir (IDV) in HIV-infected subjects with prior nucleoside analog experience. HIV Clin Trials. 2008 Jan-Feb;9(1):11-25. doi: 10.1310/hct0901-11. PMID 18215978